CLINICAL TRIAL: NCT00297700
Title: Implementing Tobacco Control in Dental Practice
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 5R01DA017974 (NIH)
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2006-07

CONDITIONS: Smoking
Keywords: Smoking; Dental; Cessation; Prevention; Control; Quitline; 5A-Model; Cost-effective
MeSH Terms: conditions — Smoking

INTERVENTIONS:
Behavioral: Active referral

SUMMARY:
Our goal is to test a dentist-hygienist team intervention to help dental patients quit smoking and determine if it can be effectively and cost-effectively implemented and sustained.

Staff in half of the HMO's 14 large dental facilities will be trained to provide brief cessation advice and assistance and to encourage smokers to talk by phone with a tobacco counselor before they leave the dental office. Phone counselors will provide brief counseling, assess stage, and offer a full list of cessation services. The Active Referral intervention strategy is both practical and innovative, as it takes advantage of available resources; efficiently distributes intervention activities between dentists, hygienists, and counseling specialists; and could be delivered in individual, small, or large dental practices. This intervention is provided as part of routine care to all patients seen for annual dental and periodontal exams.Consented patients will receive a short phone survey shortly after the exam to assess smoking status, satisfaction with delivery of support services,and satisfaction with intervention. Consented patients in treatment and control facilities will be surveyed by phone at one year to re-assess smoking status and satisfaction with services.

DETAILED DESCRIPTION:
The purpose of this behavioral effectiveness trial is to test the feasibility, effectiveness, cost-effectiveness, and sustainability of a team approach for delivering smoking cessation assistance to interested smokers seen within a single well-integrated group-model dental HMO. We and others have already demonstrated the efficacy of the 5-A model in medical and hospital clinical settings. The need now is to show that a practical and innovative team approach with a centralized tobacco quitline component 1) can be disseminated throughout dental care offices; 2) can be effectively and consistently delivered by dentists and hygienists; 3)can be maintained over time, and 4) will have a positive and cost-effective impact on patient smoking-cessation rates.

The HMO's 14 dental care offices will be randomly assigned to usual care or a Assisted Referral condition. In the Referral condition, dentists and hygienists will be trained to, as part of routine annual dental exams, assess, advise, and connect interested tobacco users by phone to a professionally staffed centralized tobacco quitline. If patients prefer, dental staff will have quitline staff call the patients back at a more convenient time. Quitline staff will offer brief counseling and assessment and a full menu of cessation services, including multi-session telephone and face-to-face programs and medications. The intervention will be provided as a part of routine care to all adult patients receiving annual general dental or periodontal exams.

Primary and secondary outcome measure. The primary hypothesis is that treatment will increase the probability of 30-day sustained cessation from all forms of tobacco, as reported by randomly selected patients one year after the initial clinic visit. Other secondary follow-up measures will include one-week and 6-month point prevalence at one year, stage of change, quit attempts during the year, and smoking rate among continuing smokers.

CHR research staff will survey a random sample of 2,800 consenting adult cigarette smokers in both Referral and Usual Care facilities shortly after their visits to assess rates of advice and referral, satisfaction, and other process measures. Patients will be sampled throughout a 15-month period to assess sustainability of the staff's efforts. Consenting patients will be resurveyed after one year to assess smoking cessation outcomes. Patients seen by dentists or hygienists who routinely practice in multiple facilities will be excluded to minimize contamination.

The Kaiser Permanente Dental Care Program (KPDCP) is a well-integrated single-group dental HMO with a unified administrative structure. KPDCP and the Kaiser Permanente Center for Health Research (CHR) are both divisions within a single institution- Kaiser Permanente Northwest. The dental program has 14 clinical facilities in the Vancouver, Washington; Portland, Oregon; and Salem, Oregon service areas. The dental plan's aim is to implement the tobacco control program as a permanent change in the routine care that is delivered to all patients throughout all facilities. In order to evaluate the change process and the impact of the program, however, they will stagger the rollout of the quality improvement effort with half of the facilities randomly assigned to begin during phase I and the remainder to start later once follow-up is complete.

While multiple clinics will offer advice and referral options to smokers, research staff at only one data collection site (i.e., CHR) will carry out all study recruitment, consent, and data collection activities as part of the post-visit and annual follow-up surveys. Because CHR is the only data collection site for study subjects, and the fact that we are all part of a single well-integrated organization operating under a single IRB, we view this as a single-site study.

Projected timeline. The first nine months of the project will be devoted to planning, development and testing the web intervention and final telephone counseling protocol, and piloting all aspects of the identification, recruitment, assessment, and intervention components of the study. Recruitment will begin shortly before year 2.

Target population distribution. The target population is 52% women, 15.9% nonwhite or mixed race, and 7.4% Hispanic.

Data acquisition and entry. Random samples of smoking patients seen for annual general dental or periodontal exams will be called to complete a short "Current Visit Survey" shortly after their visits. We will randomly select up to 4,000 smoking patients (approximately 285 per facility) to contact. We expect to achieve a minimum response rate of 70%, based on a 76% response rate achieved using this same procedure with patients seen for routine medical visits (Hollis, 2000b). A 70% response rate will yield an estimated 2,800 respondents (200 per facility).

Data analysis. Because clinics rather than patients are the unit of randomization, adjustments for the intra clinic correlation will be necessary for all treatment comparisons. The primary outcome analysis is based on the mixed effects logit model: logitY i:k:l = M +Cl +G k:l +e i:k:l (1)

The adjusted mixed effects logit model will also test for differences between the early and sustained effects of program implementation on tobacco quit rates by including a member-level time covariate (T i:k:l) and an interaction term between time and intervention effect (Cl). A significant interaction term indicates that the early and late intervention effects differ.

Delivery of the intervention components (e.g., asking, advising, and referring smokers) will be assessed primarily by analysis of the patient's reports on the post-visit phone survey they will receive shortly after the visit and the one-year follow-up phone survey. Fields in the computerized dental record will provide another somewhat limited source of information on rates of asking, advising, and referring smokers.

ELIGIBILITY:
Inclusion Criteria:

* Kaiser Permanente (KP)member
* 18 years of age or older
* Receiving routine primary care in KP dental offices
* Tobacco user at time of routine dental visit

Exclusion Criteria:

* Non-KP member
* Less than 18 years or age
* Non-tobacco user

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2800
Dates: Start 2004-05; Study Completion 2007-04

PRIMARY OUTCOMES:
Tobacco-cessation rates (30-day point prevalence) at one year.

SECONDARY OUTCOMES:
Process measures (e.g., 5As, and referrals)
Stage of change progression
Program costs

CONTACTS AND LOCATIONS:
Overall Officials: Jack F. Hollis, Ph.D., Principal Investigator — Kaiser Permanente Foundation Hospitals/ Center for Health Research
Locations (1):
- Center for Health Research, Portland, Oregon, United States

REFERENCES:
- [Background] Albert D, Ward A, Ahluwalia K, Sadowsky D. Addressing tobacco in managed care: a survey of dentists' knowledge, attitudes, and behaviors. Am J Public Health. 2002 Jun;92(6):997-1001. doi: 10.2105/ajph.92.6.997. PMID 12036795
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Bergstrom J, Eliasson S, Dock J. Exposure to tobacco smoking and periodontal health. J Clin Periodontol. 2000 Jan;27(1):61-8. doi: 10.1034/j.1600-051x.2000.027001061.x. PMID 10674963
- [Background] Bracht, N., Kingsbury, L. & Rissel L. A Five stage Community Organization Model for Health Promotion. In Bracht, N (Ed.). Health Promotion at the Community Level. International Educational and Professional Publisher. Thousand Oaks, California: SAGE Publications; 1999, pp. 83-104.
- [Background] Brothwell DJ. Should the use of smoking cessation products be promoted by dental offices? An evidence-based report. J Can Dent Assoc. 2001 Mar;67(3):149-55. PMID 11282035
- [Background] Campbell HS, Sletten M, Petty T. Patient perceptions of tobacco cessation services in dental offices. J Am Dent Assoc. 1999 Feb;130(2):219-26. doi: 10.14219/jada.archive.1999.0171. PMID 10036845
- [Background] Centers for Disease Control and Prevention (CDC). Annual smoking-attributable mortality, years of potential life lost, and economic costs--United States, 1995-1999. MMWR Morb Mortal Wkly Rep. 2002 Apr 12;51(14):300-3. PMID 12002168
- [Background] Coffield AB, Maciosek MV, McGinnis JM, Harris JR, Caldwell MB, Teutsch SM, Atkins D, Richland JH, Haddix A. Priorities among recommended clinical preventive services. Am J Prev Med. 2001 Jul;21(1):1-9. doi: 10.1016/s0749-3797(01)00308-7. PMID 11418251
- [Background] Cohen SJ, Stookey GK, Katz BP, Drook CA, Christen AG. Helping smokers quit: a randomized controlled trial with private practice dentists. J Am Dent Assoc. 1989 Jan;118(1):41-5. doi: 10.14219/jada.archive.1989.0018. PMID 2913103
- [Background] Cromwell J, Bartosch WJ, Fiore MC, Hasselblad V, Baker T. Cost-effectiveness of the clinical practice recommendations in the AHCPR guideline for smoking cessation. Agency for Health Care Policy and Research. JAMA. 1997 Dec 3;278(21):1759-66. PMID 9388153
- [Background] Cummings SR, Rubin SM, Oster G. The cost-effectiveness of counseling smokers to quit. JAMA. 1989 Jan 6;261(1):75-9. PMID 2491762
- [Background] Curry SJ. Organizational interventions to encourage guideline implementation. Chest. 2000 Aug;118(2 Suppl):40S-46S. doi: 10.1378/chest.118.2_suppl.40s. PMID 10939998
- [Background] Drummond MF, O'Brien B, Stoddart GL, Torrance GW. Methods for the Economic Evaluation of Health Care Programmes, 2nd ed. Oxford: Oxford University Press, 1997.
- [Background] Eddy DM, David Eddy ranks the tests. Harvard Health Letters 1992; July Supplement:10-11.
- [Background] Farnham PG, Haddix AC. Study design. In: Haddix AC, Teutsch, Corso PS, eds. Prevention Effectiveness. New York: Oxford University Press, 2003, pp. 11-27.
- [Background] Fichtenberg CM, Glantz SA. Association of the California Tobacco Control Program with declines in cigarette consumption and mortality from heart disease. N Engl J Med. 2000 Dec 14;343(24):1772-7. doi: 10.1056/NEJM200012143432406. PMID 11114317
- [Background] Fiore MC. AHCPR smoking cessation guideline: a fundamental review. Tob Control. 1997;6 Suppl 1:S4-8. No abstract available. PMID 9396115
- [Background] Fiore MC, Bailey WC, Cohen SJ, et al. Clinical Practice Guideline Smoking Cessation. Rockville, MD: U.S. Department of Health and Human Services; 1996.
- [Background] Fiore MC, Bailey WC, Cohen SJ, et al. Treating Tobacco Use and Dependence: A Clinical Practice Guideline. Rockville, MD: U.S. Department of Health and Human Services; 2000. Available at www.surgeongeneral.gov/tobacco
- [Background] Glasgow RE, Hollis JF, McRae SG, Lando HA, LaChance P. Providing an integrated program of low intensity tobacco cessation services in a health maintenance organization. Health Educ Res. 1991 Mar;6(1):87-99. doi: 10.1093/her/6.1.87. PMID 10148728
- [Background] Glasgow RE, Mullooly JP, Vogt TM, Stevens VJ, Lichtenstein E, Hollis JF, Lando HA, Severson HH, Pearson KA, Vogt MR. Biochemical validation of smoking status: pros, cons, and data from four low-intensity intervention trials. Addict Behav. 1993 Sep-Oct;18(5):511-27. doi: 10.1016/0306-4603(93)90068-k. PMID 8310871
- [Background] Gordon JS, Severson HH. Tobacco cessation through dental office settings. J Dent Educ. 2001 Apr;65(4):354-63. PMID 11336121
- [Background] Grimshaw JM, Shirran L, Thomas R, Mowatt G, Fraser C, Bero L, Grilli R, Harvey E, Oxman A, O'Brien MA. Changing provider behavior: an overview of systematic reviews of interventions. Med Care. 2001 Aug;39(8 Suppl 2):II2-45. PMID 11583120
- [Background] Haddix AC, Teutsch, Corso PS, eds. Prevention Effectiveness. New York: Oxford University Press, 2003.
- [Background] Hall SM, Delucchi KL, Velicer WF, Kahler CW, Ranger-Moore J, Hedeker D, Tsoh JY, Niaura R. Statistical analysis of randomized trials in tobacco treatment: longitudinal designs with dichotomous outcome. Nicotine Tob Res. 2001 Aug;3(3):193-202. doi: 10.1080/14622200110050411. PMID 11506764
- [Background] Hollis JF. Population impact of clinician efforts to reduce tobacco use. National Cancer Institute. Population Based Smoking Cessation: Proceedings of a Conference on What Works to Influence Cessation in the General Population. Smoking and Tobacco Control Monograph No. 10. Bethesda, MD: U.S. Department of Health and Human Services, National Institutes of Health, National Cancer Institute, NIH Pub. No. 00-4892, November 2000a.
- [Background] Hollis JF, Bills R, Whitlock E, Stevens VJ, Mullooly J, Lichtenstein E. Implementing tobacco interventions in the real world of managed care. Tob Control. 2000;9 Suppl 1(Suppl 1):I18-24. doi: 10.1136/tc.9.suppl_1.i18. No abstract available. PMID 10688926
- [Background] Hollis JF, Lichtenstein E, Mount K, Vogt TM, Stevens VJ. Nurse-assisted smoking counseling in medical settings: minimizing demands on physicians. Prev Med. 1991 Jul;20(4):497-507. doi: 10.1016/0091-7435(91)90047-8. PMID 1871078
- [Background] Hollis JF, Vogt TM, Stevens VJ, Biglan A, Severson H, Lichtenstein E. The tobacco reduction and cancer control (TRACC) program: Team approaches to counseling in medical and dental settings. In: Burns DM, Gritz ER, eds., Tobacco and the Clinician: Interventions for Medical and Dental Practice. National Cancer Institute, Monograph 5, NIH Publication No. 94-3693, 1994.
- [Background] Hollis JF, Lichtenstein E, Vogt TM, Stevens VJ, Biglan A. Nurse-assisted counseling for smokers in primary care. Ann Intern Med. 1993 Apr 1;118(7):521-5. doi: 10.7326/0003-4819-118-7-199304010-00006. PMID 8442622
- [Background] Kiefe CI, Allison JJ, Williams OD, Person SD, Weaver MT, Weissman NW. Improving quality improvement using achievable benchmarks for physician feedback: a randomized controlled trial. JAMA. 2001 Jun 13;285(22):2871-9. doi: 10.1001/jama.285.22.2871. PMID 11401608
- [Background] Kottke TE, Battista RN, DeFriese GH, Brekke ML. Attributes of successful smoking cessation interventions in medical practice. A meta-analysis of 39 controlled trials. JAMA. 1988 May 20;259(19):2883-9. doi: 10.1001/jama.259.19.2883. PMID 3367456
- [Background] Leininger LS, Finn L, Dickey L, Dietrich AJ, Foxhall L, Garr D, Stewart B, Wender R. An office system for organizing preventive services: a report by the American Cancer Society Advisory Group on Preventive Health Care Reminder Systems. Arch Fam Med. 1996 Feb;5(2):108-15. doi: 10.1001/archfami.5.2.108. PMID 8601207
- [Background] Lichtenstein E, Hollis JF, Severson HH, Stevens VJ, Vogt TM, Glasgow RE, Andrews JA. Tobacco cessation interventions in health care settings: rationale, model, outcomes. Addict Behav. 1996 Nov-Dec;21(6):709-20. doi: 10.1016/0306-4603(96)00030-5. PMID 8904937
- [Background] Lichtenstein E, Hollis J. Patient referral to a smoking cessation program: who follows through? J Fam Pract. 1992 Jun;34(6):739-44. PMID 1593248
- [Background] Bernard HR, Ryan GW. Text analysis: Qualitative and quantitative methods. In: Bernard HR, editor. Handbook of Methods in Cultural Anthropology. Walnut Creek, CA: AltaMira Press; 1998.
- [Background] Little SJ, Stevens VJ, Severson HH, Lichtenstein E. Effective smokeless tobacco intervention for dental hygiene patients. J Dent Hyg. 1992 May;66(4):185-90. PMID 1625002
- [Background] Little SJ, Stevens VJ. Dental hygiene's role in reducing tobacco use. A literature review and recommendations for action. J Dent Hyg. 1991 Sep;65(7):346-50. No abstract available. PMID 1819632
- [Background] Martin LM, Bouquot JE, Wingo PA, Heath CW Jr. Cancer prevention in the dental practice: oral cancer screening and tobacco cessation advice. J Public Health Dent. 1996 Fall;56(6):336-40. doi: 10.1111/j.1752-7325.1996.tb02461.x. PMID 9089529
- [Background] McAfee T, Sofian NS, Wilson J, Hindmarsh M. The role of tobacco intervention in population-based health care: a case study. Am J Prev Med. 1998 Apr;14(3 Suppl):46-52. doi: 10.1016/s0749-3797(97)00051-2. PMID 9566937
- [Background] Miller WL, Crabtree BF. Qualitative analysis: how to begin making sense. Fam Pract Res J. 1994 Sep;14(3):289-97. PMID 7976480
- [Background] Miller WR, Rollnick S. Motivational Interviewing. New York, NY: The Guilford Press; 1991.
- [Background] Morgan DL. The Focus Group Guidebook. Thousand Oaks, CA: Sage; 1998.
- [Background] Murray DM. Design and Analysis of Group Randomized Trials. Oxford, NY: The Oxford University Press; 1998.
- [Background] Thomson O'Brien MA, Oxman AD, Haynes RB, Davis DA, Freemantle N, Harvey EL. Local opinion leaders: effects on professional practice and health care outcomes. Cochrane Database Syst Rev. 2000;(2):CD000125. doi: 10.1002/14651858.CD000125. PMID 10796491
- [Background] Ockene JK. Smoking intervention: the expanding role of the physician. Am J Public Health. 1987 Jul;77(7):782-3. doi: 10.2105/ajph.77.7.782. No abstract available. PMID 3592029
- [Background] Ockene JK. Physician-delivered interventions for smoking cessation: strategies for increasing effectiveness. Prev Med. 1987 Sep;16(5):723-37. doi: 10.1016/0091-7435(87)90054-5. PMID 3317393
- [Background] Orleans CT, George LK, Houpt JL, Brodie KH. Health promotion in primary care: a survey of U.S. family practitioners. Prev Med. 1985 Sep;14(5):636-47. doi: 10.1016/0091-7435(85)90083-0. PMID 4070193
- [Background] Orleans CT, Schoenbach VJ, Wagner EH, Quade D, Salmon MA, Pearson DC, Fiedler J, Porter CQ, Kaplan BH. Self-help quit smoking interventions: effects of self-help materials, social support instructions, and telephone counseling. J Consult Clin Psychol. 1991 Jun;59(3):439-48. doi: 10.1037//0022-006x.59.3.439. PMID 2071729
- [Background] Oxman AD, Thomson MA, Davis DA, Haynes RB. No magic bullets: a systematic review of 102 trials of interventions to improve professional practice. CMAJ. 1995 Nov 15;153(10):1423-31. PMID 7585368
- [Background] Pederson LL. Compliance with physician advice to quit smoking: a review of the literature. Prev Med. 1982 Jan;11(1):71-84. doi: 10.1016/0091-7435(82)90006-8. No abstract available. PMID 7079248
- [Background] Prochaska JO, Velicer WF. The transtheoretical model of health behavior change. Am J Health Promot. 1997 Sep-Oct;12(1):38-48. doi: 10.4278/0890-1171-12.1.38. PMID 10170434
- [Background] Prochaska JO, DiClemente CC. Stages and processes of self-change of smoking: toward an integrative model of change. J Consult Clin Psychol. 1983 Jun;51(3):390-5. doi: 10.1037//0022-006x.51.3.390. No abstract available. PMID 6863699
- [Background] Prochaska JO, DiClemente CC, Velicer WF, Rossi JS. Criticisms and concerns of the transtheoretical model in light of recent research. Br J Addict. 1992 Jun;87(6):825-8; discussion 833-5. doi: 10.1111/j.1360-0443.1992.tb01973.x. No abstract available. PMID 1525523
- [Background] Rigotti NA, Quinn VP, Stevens VJ, Solberg LI, Hollis JF, Rosenthal AC, Zapka JG, France E, Gordon N, Smith S, Monroe M. Tobacco-control policies in 11 leading managed care organizations: progress and challenges. Eff Clin Pract. 2002 May-Jun;5(3):130-6. PMID 12088292
- [Background] Rost K, Burnam MA, Smith GR. Development of screeners for depressive disorders and substance disorder history. Med Care. 1993 Mar;31(3):189-200. doi: 10.1097/00005650-199303000-00001. PMID 8450677
- [Background] Severson HH, Andrews JA, Lichtenstein E, Gordon JS, Barckley MF. Using the hygiene visit to deliver a tobacco cessation program: results of a randomized clinical trial. J Am Dent Assoc. 1998 Jul;129(7):993-9. doi: 10.14219/jada.archive.1998.0353. PMID 9685764
- [Background] Silagy C, Lancaster T, Gray S, Fowler G. Effectiveness of training health professionals to provide smoking cessation interventions: systematic review of randomised controlled trials. Qual Health Care. 1994 Dec;3(4):193-8. doi: 10.1136/qshc.3.4.193. PMID 10140233
- [Background] Solas V.3.0. Cork, Ireland; Statistical Solutions Ltd., 2001.
- [Background] Solberg LI, Kottke TE, Conn SA, Brekke ML, Calomeni CA, Conboy KS. Delivering clinical preventive services is a systems problem. Ann Behav Med. 1997 Summer;19(3):271-8. doi: 10.1007/BF02892291. PMID 9603701
- [Background] SRNT Subcommittee on Biochemical Verification. Biochemical verification of tobacco use and cessation. Nicotine Tob Res. 2002 May;4(2):149-59. doi: 10.1080/14622200210123581. No abstract available. PMID 12028847
- [Background] Stevens VJ, Severson H, Lichtenstein E, Little SJ, Leben J. Making the most of a teachable moment: a smokeless-tobacco cessation intervention in the dental office. Am J Public Health. 1995 Feb;85(2):231-5. doi: 10.2105/ajph.85.2.231. PMID 7856783
- [Background] Stevens VJ, Hollis JF. Preventing smoking relapse, using an individually tailored skills-training technique. J Consult Clin Psychol. 1989 Jun;57(3):420-4. doi: 10.1037//0022-006x.57.3.420. PMID 2738215
- [Background] Stevens VJ, Glasgow RE, Hollis JF, Lichtenstein E, Vogt TM. A smoking-cessation intervention for hospital patients. Med Care. 1993 Jan;31(1):65-72. doi: 10.1097/00005650-199301000-00005. PMID 8417271
- [Background] Thun MJ, Day-Lally C, Myers DG, Calle EE, Flanders WD, Zhu B-P, Namboodiri MM, Heath CW Jr. Trends in tobacco smoking and mortalityfrom cigarette use in Cancer Prevention Studies I (1959 through 1965) and II (1982 through 1988). In: Changes in Cigarette-Related Disease Risks and Their Implication for prevention and Control. National Cancer Institute, NIH Publication No. 97-4213, 1997.
- [Background] Tomar SL, Asma S. Smoking-attributable periodontitis in the United States: findings from NHANES III. National Health and Nutrition Examination Survey. J Periodontol. 2000 May;71(5):743-51. doi: 10.1902/jop.2000.71.5.743. PMID 10872955
- [Background] Tomar SL, Winn DM. Chewing tobacco use and dental caries among U.S. men. J Am Dent Assoc. 1999 Nov;130(11):1601-10. doi: 10.14219/jada.archive.1999.0099. PMID 10573940
- [Background] Tomar SL. Dentistry's role in tobacco control. J Am Dent Assoc. 2001 Nov;132 Suppl:30S-35S. doi: 10.14219/jada.archive.2001.0386. PMID 11803650
- [Background] U.S. Department of Health and Human Services. The health benefits of smoking cessation (DHHS Publication No. (CDC) 90-8416). Washington DC: U.S. Department of Health and Human Services, Public Health Service, Centers for Disease Control, 1990.
- [Background] Velicer WF, Prochaska JO, Rossi JS, Snow MG. Assessing outcome in smoking cessation studies. Psychol Bull. 1992 Jan;111(1):23-41. doi: 10.1037/0033-2909.111.1.23. PMID 1539088
- [Background] Vogt TM, Lichtenstein E, Ary D, Biglan A, Danielson R, Glasgow RE, Hollis JF, Hornbrook MC, Lando H, Severson H, Stevens V. Integrating tobacco intervention into a health maintenance organization: The TRACC Program. Health Education Research 1989; 4:125-135.
- [Background] Warner KE, Warner PA. Is an ounce of prevention worth a pound of cure? Disease prevention in health care reform. J Ambul Care Manage. 1993 Oct;16(4):38-49. doi: 10.1097/00004479-199310000-00007. No abstract available. PMID 10128416
- [Background] Warner KE. Cost effectiveness of smoking-cessation therapies. Interpretation of the evidence-and implications for coverage. Pharmacoeconomics. 1997 Jun;11(6):538-49. doi: 10.2165/00019053-199711060-00003. PMID 10168094
- [Background] Weinstein MC, Siegel JE, Gold MR, Kamlet MS, Russell LB. Recommendations of the Panel on Cost-effectiveness in Health and Medicine. JAMA. 1996 Oct 16;276(15):1253-8. PMID 8849754
- [Derived] Holliday R, Hong B, McColl E, Livingstone-Banks J, Preshaw PM. Interventions for tobacco cessation delivered by dental professionals. Cochrane Database Syst Rev. 2021 Feb 19;2(2):CD005084. doi: 10.1002/14651858.CD005084.pub4. PMID 33605440